CLINICAL TRIAL: NCT01662232
Title: The Role of EGCG in Different Application Forms on Flow-mediated Dilation in Healthy Volunteers
Brief Title: Improvement of Endothelial Function by EGCG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Mario Lorenz, PhD, PhD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Char-EGCG-FMD
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases
Keywords: Green tea; EGCG; Cardiovascular diseases; Endothelial function; Flow-mediated dilation
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Green tea beverage (Active Comparator): 200 mg EGCG as green tea beverage.
  Interventions: Dietary Supplement: Green tea beverage
- Green tea extract (Active Comparator): 200 mg EGCG as green tea extract and same volume water as for tea beverage.
  Interventions: Dietary Supplement: Green tea extract
- Epigallocatechin-3-gallate (EGCG) (Active Comparator): 200 mg EGCG and same volume water as for tea beverage.
  Interventions: Dietary Supplement: EGCG
- Placebo (Water) (Placebo Comparator): Same volume water as for all intervention arms.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Green tea beverage
  Arms: Green tea beverage
Dietary Supplement: Green tea extract
  Arms: Green tea extract
Dietary Supplement: EGCG
  Arms: Epigallocatechin-3-gallate (EGCG)
Other: Placebo
  Arms: Placebo (Water)

SUMMARY:
Cardiovascular diseases are a major cause of morbidity and mortality worldwide. Impaired endothelial function (assessed as flow-mediated dilation) represents an early marker for later cardiovascular events. Epidemiological and experimental studies suggest that consumption of tea is associated with lower progression of atherosclerosis and reduced cardiovascular mortality.

Tea contains high amounts of polyphenols with important biological activities. The green tea catechin epigallocatechin-3-gallate (EGCG) is the most potent physiologically active compound in vitro. However, little is known about its contribution to beneficial effects of tea in vivo.

In this crossover study the impact of a single dose of EGCG applied in different forms (green tea beverage, green tea extract and EGCG) on flow-mediated dilation is investigated in healthy volunteers two hours after ingestion. The amount of EGCG (200 mg) corresponds to appr. 0.5 L of green tea. The results of the study will elucidate the contribution of EGCG in cardiovascular protective effects of green tea in vivo. The outcomes will provide insights about the role of EGCG in different application forms to improvements of endothelial function in humans.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteers
* 20-50 years
* BMI < 27 kg/m2
* Cholesterol < 240 mg/dl

Exclusion Criteria:

* Diabetes mellitus
* Hypertension
* Conditions with impaired endothelial function
* Smoking
* Regular drug use
* Alcohol abuse
* Regular tea drinkers

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation of the arteria brachialis | 2 hours after ingestion
  Change in flow-mediated dilation (in %) of the arteria brachialis after a single dose of 200 mg EGCG either as green tea beverage, green tea extract or EGCG is assessed by vascular ultrasound.

SECONDARY OUTCOMES:
Agonist-induced platelet aggregation in vitro | 2 hours after ingestion
  Blood is drawn two hours after consumption and the effects on in vitro agonist-induced platelet aggregation after a single dose of 200 mg EGCG either as green tea beverage, green tea extract or EGCG are measured.
Determination of plasma tea polyphenol levels | 2 hours after ingestion
  Blood is drawn two hours after consumption and plasma concentrations of tea polyphenols are measured after a single dose of 200 mg EGCG either as green tea beverage, green tea extract or EGCG by HPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Lorenz, PhD, Principal Investigator — Department of Cardiology and Angiology, Campus Mitte, Charité University Medicine Berlin, Germany
Locations (1):
- Department of Cardiology and Angiology, Campus Mitte, Charité University Medicine Berlin, Berlin, State of Berlin, Germany